CLINICAL TRIAL: NCT00307450
Title: Efficacy and Safety of Levetiracetam Versus Placebo on Levodopa-induced Dyskinesias in Advanced Parkinson's Disease (LeLeDys Study) - A Multicenter, Randomized, Stratified, Double-blinded, Placebo-controlled Phase IV Study
Brief Title: Efficacy and Safety of Levetiracetam Versus Placebo on Levodopa-induced Dyskinesias in Advanced Parkinson's Disease
Acronym: LeLeDys
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: UCB Pharma GmbH (Industry)
Responsible Party: Prof. Dr. med. Alexander Storch, Dresden University of Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TUD-LELEDY-007; Ethic board no.: EK10012006; EUDRAC no.: 2005-005940-18
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Parkinson's Disease
Keywords: Dyskinesias; Parkinson's disease; Levetiracetam; Treatment
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Levetiracetam — up to 200 mg per day in two dosages per day.

SUMMARY:
The study is designed to measure the efficacy and safety of levetiracetam on levodopa-induced dyskinesias in late-stage Parkinson's disease. The patients are planned to be treated with levetiracetam (up to 2000 mg per day) or placebo for 13 weeks. Efficacy measure is the modified AIMS.

DETAILED DESCRIPTION:
The LeLeDys study is designed to determine the efficacy and safety of levetiracetam on levodopa-induced dyskinesias in advanced Parkinson's disease.

The design is a multicenter, randomized, stratified, double-blinded, placebo-controlled phase IV study design.

The hypothesis is that levetiracetam is able to reduce duration and severity of levodopa-induced dyskinesias in Parkinson's disease.

The patients are planned to be treated with levetiracetam (up to 2000 mg per day) or placebo for 13 weeks. Efficacy measure is the modified AIMS.

Main inclusion criteria are:

* Advanced Parkinson's disease (Hoehn & Yahr II-IV)
* Age of 30 to 80 years
* Levodopa-induced dyskinesias of at least 25% of the waking day and with moderate disability
* Stable dosage of antiparkinson medication and/or stable deep brain stimulation parameters for at least 4 week prior inclusion
* Written informed consent

Main exclusion criteria are:

* Atypical parkinsonian syndromes
* Treatment with antipsychotics
* Epilepsia or seizure in the history
* Deep brain stimulation other than DBS in STN
* Pregnant or lactating women
* Severe dementia

Methods:

* Primary outcome measure is the modified AIMS
* Secondary outcome measures include UPDRS, safety, patient day record

Study medication:

* Levetiracetam (upt to 2000 mg / day)
* Matched Placebo

ELIGIBILITY:
Inclusion Criteria:

* Advanced Parkinson's disease (Hoehn & Yahr II-IV)
* Age of 30 to 80 years
* Levodopa-induced dyskinesias of at least 25% of the waking day and with moderate disability
* Stable dosage of antiparkinson medication and/or stable deep brain stimulation parameters for at least 4 week prior inclusion
* Written informed consent

Exclusion Criteria:

* Atypical parkinsonian syndromes
* Treatment with antipsychotics
* Epilepsia or seizure in the history
* Deep brain stimulation other than DBS in STN
* Pregnant or lactating women
* Severe dementia

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2006-03; Primary Completion 2009-03 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Modified AIMS | 11 weeks
UPDRS items 32 & 33 | 11 weeks

SECONDARY OUTCOMES:
UPDRS | 11 weeks
Schwab & England scale | 11 weeks
Hoehn & Yahr scale | 11 weeks
GCI | 11 weeks
Patient day record | 11 weeks
Epsworth sleep scale | 11 weeks
Levodopa challenge test | 11 weeks
Safety measures | 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Storch, M, Principal Investigator — Technical University of Dresden
Locations (2):
- Germany (2):
  - Department of Neurology at the Technical University of Dresden, Dresden
  - Department of Neurology at the University of Leipzig, Leipzig

REFERENCES:
- See also: Related Info — http://www.neuro.med.tu-dresden.de